CLINICAL TRIAL: NCT01153828
Title: Pharmacovigilence for Retapamulin: Age-stratified Monitoring of Prescribed Use in the European Union
Brief Title: EU PV for Retapamulin-Prescribing
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113149
Record Dates: First submitted 2010-05-13; First posted 2010-06-30 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-05

CONDITIONS: Impetigo
Keywords: Altargo; Bactroban; Fucidin; Fusidic acid; Mupirocin; topical; Retapamulin; United Kingdom
MeSH Terms: conditions — Impetigo | interventions — retapamulin; Mupirocin; Fusidic Acid

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- (1) Age <9 months: Age at time of prescription was <9 months
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin; Drug: Co-prescription of retapamulin and topical fusidic acid
- (2) 9 months to 6 years: Age at time of prescription was 9 months to 6 years
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin; Drug: Co-prescription of retapamulin and topical fusidic acid
- (3) 7 years to 18 years: Age at time of prescription was 7 years to 18 years
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin; Drug: Co-prescription of retapamulin and topical fusidic acid
- (4) 19 to 65 years: Age at time of prescription was 19 to 65 years
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin; Drug: Co-prescription of retapamulin and topical fusidic acid
- (5) 66 years and older: Age at time of prescription was 66 years and older
  Interventions: Drug: Retapamulin; Drug: Co-prescription of retapamulin and topical mupirocin; Drug: Co-prescription of retapamulin and topical fusidic acid

INTERVENTIONS:
Drug: Retapamulin — Prescription for retapamulin
Drug: Co-prescription of retapamulin and topical mupirocin — Same day prescriptions for retapamulin and topical mupirocin
Drug: Co-prescription of retapamulin and topical fusidic acid — Same day prescription for retapamulin and fusidic acid.

SUMMARY:
Retapamulin, a topical pleuromutilin antibiotic, is the first in a new class of topical antibiotics approved for human use. In the European Union (EU), retapamulin is approved for the treatment of impetigo and secondarily-infected traumatic lesions in persons nine or more months of age. This study is designed to examine retapamulin use in the pediatric population less than nine months of age. We will conduct a five-year assessment of prescriptions for retapamulin using the General Practice Research Database. For each year of reporting, the observed frequencies of prescriptions of retapamulin, with or without same-day co-prescriptions of topical mupirocin or fusidic acid, will be identified. The five-year reporting period will include five years of distinct, non-overlapping, non-cumulative prescription use of first exposure to retapamulin, with or without same-day co-prescription of topical mupirocin or fusidic acid.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of all registered "research standard" patients on GPRD, as evaluated annually for five years. For each year of observation, the denominator of persons will be patients registered for at least one month during the prior calendar year. Hence, the five-year reporting period for distinct, non-overlapping, non-cumulative prescription use and will categorize persons by date of birth (mm/dd/year).

Exclusion Criteria:

* Enrollment in GPRD of less than one month duration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The GPRD contains detailed information for a sample of patients from representative general practices throughout the United Kingdom. Patient data included in the GPRD were drawn from the computer systems used by general practitioners to maintain the clinical records within their practices and contain all records deemed relevant to patient care. Prescriptions of Altabax, Altargo, Mupirocin and Fucidin will be captured.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Prescription for retapamulin | First prescription in database for each calendar year between January 2007 and December 2011

SECONDARY OUTCOMES:
Co-prescription of retapamulin and topical mupirocin | First same-day prescriptions for both medicines in database for each calendar year between January 2007 and December 2011
Co-prescription of retapamulin and topical fusidic acid | First same-day prescriptons for both medicines in database for each calendar year between January 2007 and December 2011

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline